CLINICAL TRIAL: NCT03221010
Title: Evaluation of the Effectiveness of the Motivational Interviewing in the Cessation of Smoking in Groups in Primary Health Care Services: a Community Clinical Trial
Brief Title: Use of the Motivational Interviewing in the Treatment of Smokers in Groups in Primary Health Care
Acronym: MITG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Daniel Demétrio Faustino da Silva, Dentist, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HNSC-Tobacco Groups
Record Dates: First submitted 2017-07-16; First posted 2017-07-18 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Smoking, Tobacco; Smoking Cessation
Keywords: Smoking; Smoking cessation; Motivational Interviewing; Primary health care; Randomized clinical trial
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation; Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Intervention Group: in this group, composed of 6 randomized Basic Health Units, the professionals who coordinate the smoking groups will receive the training for the use of the Motivational Interviewing as an additional resource to the work of motivation and cognitive-behavioral approach usually performed in the groups, however , With an approach based on Motivational Interviewing.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Traditional cognitive-behavioral approach
- Traditional cognitive-behavioral approach (Active Comparator): Control Group: in this group composed of the remaining 6 Randomized Basic Health Units, professionals will use only the traditional cognitive-behavioral approach advocated by the Brazilian Ministry of Health's smoking program.
  Interventions: Behavioral: Traditional cognitive-behavioral approach

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interview (MI) is a person-centered, communicative method whose purpose is to work and increase the user's motivation for behavior change.
  Arms: Motivational Interviewing
Behavioral: Traditional cognitive-behavioral approach — This approach aims to combine cognitive interventions in the training of behavioral skills in patients, developing strategies to cope with the problem and detecting situations of risk, mobilizing the subject for his own process of change. Helps correct cognitive dysfunctions and behavioral changes in specific situations.
  Other Names: cognitive-behavioral approach

SUMMARY:
The objective of this study is to evaluate the efficacy of Motivational Interview (MI) on the smoking cessation rates of the smoking groups performed by the primary care teams of the Conceição Hospitalar Group, Porto Alegre, Brasil, and also whether there is an increase in the completion rate of the groups.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable death and a major public health problem worldwide. Primary health care is a strategic setting in the treatment of this problem. The objective of this study is to evaluate the efficacy of Motivational Interview (MI) on the smoking cessation rates of the smoking groups performed by the primary care teams of the Conceição Hospitalar Group, Porto Alegre, Brasil, and also whether there is an increase in the completion rate of the groups. Methodology: A randomized community trial was carried out in the 12 units of this service, starting in July 2016, with randomization by cluster, where the intervention group received an 8-hour training in MI in order to associate the technique with the conventional approach, while the units of the control group used only the conventional approach.

ELIGIBILITY:
Inclusion Criteria:

* Smokers.
* Participate in group smoking treatment.

Exclusion Criteria:

* Missing more than two sessions of the smoking group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | thirty days
  Smoking cessation rate

CONTACTS AND LOCATIONS:
Locations (1):
- Nossa Senhora da Conceição Hospital, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No